CLINICAL TRIAL: NCT01619540
Title: Study of the Valsalva Manœuvre in the Diagnosis of Left Ventricular Failure During Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: Valsalva Manœuvre in the Diagnosis of Left Ventricular Failure in Chronic Obstructive Pulmonary Disease Exacerbation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Nouira, Study of the Valsalva Manœuvre in Diagnoses of Left Ventricular Failure During Acute Exacerbation of Chronic Obstructive Pulmonary Desease, University of Monastir
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: Valsalva
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Acute Heart Failure; COPD Exacerbation
Keywords: COPD; Left Ventricular Failure; Valsalva Manoeuver
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure | interventions — Valsalva Maneuver

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- acute heart failure (Other): control arm
  Interventions: Other: Valsalva maneuver
- COPD exacerbation (Experimental): COPD exacerbation
  Interventions: Other: Valsalva maneuver

INTERVENTIONS:
Other: Valsalva maneuver

SUMMARY:
Left ventricular failure (LVF) is a common cause of acute exacerbation of chronic obstructive pulmonary disease (AECOPD).

This association is frequently underestimated with regard to the difficulty of clinical diagnosis .

The investigators expect that Valsalva Maneuver (VM) could be useful in this issue.

ELIGIBILITY:
Inclusion Criteria

* We included in this group, patients with a history (previous history) of COPD who consulted the emergency room for an exacerbation of COPD defined by a respiratory rate> 25c/min and a pH <7.35 and a PaCO2 >6 KPa.
* This group is also divided into two groups according to clinical expert assessment and the BNP value: Group1 : BNP> 400pg/ml, Group2 : BNP <400PG / ml

Exclusion Criteria:

* We excluded from this study patients with Prominent cardiac arrest
* Rhythm disorders including severe tachycardia arrhythmia
* Auricular fibrillation
* Hemodynamic instability requiring the use of vasoactive drugs and a contre indications of non invasive ventilation such us consciousness disorders with a Glasgow score <12/15,a swallowing disorder
* A significant bronchial obstruction ,the upper airway obstruction , in upper gastrointestinal bleeding in progress, an extreme obesity and Cirrhosis or cancer.
* We are also excluded patients who did not cooperate and those who refused the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
left ventricular dysfunction | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Semir, Professor, Principal Investigator — Monastir University
Locations (4):
- Tunisia (4):
  - Fattouma Bourguiba University hospital, Monastir, Monastir Governorate
  - University hospital of Moastir, Monastir, Monastir Governorate
  - University hospital of Monastir, Monastir, Monastir Governorate
  - University Hospital of Monastir, Monastir, Monstir

REFERENCES:
- [Derived] Boubaker H, Grissa MH, Debbabi H, Beltaief K, Dridi Z, Najjar MF, Bouida W, Boukef R, Marghli S, Nouira S. Value of Plethysmographic Pulse Amplitude Ratio With Valsalva Maneuver in Identifying Left Ventricular Dysfunction During COPD Exacerbation. Respir Care. 2016 Apr;61(4):439-46. doi: 10.4187/respcare.04091. Epub 2015 Dec 8. PMID 26647450